CLINICAL TRIAL: NCT02524249
Title: A Randomized Double Blind Controlled Trial of Early Versus Late Caffeine for Extremely Low Birth Weight Newborns
Brief Title: Early Versus Late Caffeine for ELBW Newborns
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Frequent protocol violations
Sponsor: Wayne State University (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Dr. Nithin Shashikanth Chouthai, Professor of Pediatrics, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1506014098
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2019-06

CONDITIONS: Bronchopulmonary Dysplasia; Apnea of Prematurity
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Apnea | interventions — Caffeine; Glucose

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early caffeine group (Active Comparator): 55 newborns will be randomized to receive caffeine within 24 hours of life. They will receive 20mg/kg IV bolus followed by IV or PO 5mg/kg daily for the next 14 days. The clinical team may decide to give PO caffeine if the newborn tolerates >75% of fluid goals by feeds.
  Interventions: Drug: Caffeine
- Late caffeine group (Placebo Comparator): 55 newborns will be randomized to receive a placebo (dextrose) in the first 24 hours of life. They will receive a 20mg/kg IV bolus followed by IV or PO 5mg/kg daily for the next 14 days. The clinical team may decide to give the placebo orally is the newborn tolerates >75% of fluid goals by feeds.
  Interventions: Drug: Placebo (dextrose)

INTERVENTIONS:
Drug: Caffeine
  Arms: Early caffeine group
Drug: Placebo (dextrose)
  Arms: Late caffeine group

SUMMARY:
Caffeine is routinely used in the management of apnea of prematurity. Extremely low birth weight (ELBW) infants are at higher risk of mortality and various neonatal morbidities such as bronchopulmonary dysplasia (BPD) for which caffeine has been shown to be beneficial in very low birth weight (VLBW) infants. The investigators' previous unpublished retrospective studies and recently published retrospective studies demonstrated that early caffeine given within 48 hours of age tended to decrease the incidence of death and BPD in ELBW newborns. Retrospective design can be biased as newborns with mild lung disease may have received caffeine early for extubation. There are several studies on pharmacodynamics and pharmacokinetics of caffeine. The data regarding cumulative dosage of caffeine, caffeine levels and BPD outcome is deficient.

Primary objective of this study is to test the hypothesis that early caffeine given within 24 hours of life will decrease incidence of mortality and BPD in ventilated ELBW newborns.

This study will also test an additional hypothesis that higher caffeine dosage and caffeine levels are associated with decreased mortality and postnatal morbidities in studied newborns.

DETAILED DESCRIPTION:
Parents will be approached either prenatally for an impending delivery of ELBW newborn or within 16 hours of birth. 90 newborns will be randomized to receive early caffeine within 24 hours of life (the "study drug") and 90 newborns will receive a placebo. Either the early caffeine (the "study drug") or placebo will be continued throughout the first 15 days of life. Newborns in the early caffeine group will receive an IV bolus of 20mg/kg followed by IV or PO 5mg/kg daily for 14 days. The clinical team can choose to give PO caffeine if the newborn tolerates >75% of fluid goals by feeds. The clinical and research teams will be blinded; neither will know whether the newborn is receiving early caffeine or placebo. The clinical team will be allowed to use open labeled caffeine as deemed medically necessary after 24 hours of receiving either the early caffeine or placebo. Often this clinical need would be at the time of extubation (peri-extubation) and comprises the "late" caffeine group, which is also the placebo group. Perinatal and postnatal clinical characteristics will be prospectively collected. Clinical team may choose to hold study drug if newborns are placed on high frequency ventilation or if they need sedation drips for surgical procedures. Two blood samples will be collected one at day 7 and one at day 14 for caffeine levels. Data safety monitoring committee will be review mortality and morbidity in each group on a quarterly basis or after recruitment of every 30 newborns whichever happens earlier.

ELIGIBILITY:
Inclusion Criteria:

* newborns with birth weight less than or equal to 1000grams and less than 28 weeks of gestation are included if intubated by 12 hours of life

Exclusion Criteria:

* newborns with known congenital malformation
* newborns whose parents refuse consent for the study
* newborns who are on high frequency ventilation and/or receiving more than 80% oxygen at 12 hours of age
* newborns deemed non-viable by the clinical team (defined as those neonates born at <24 weeks gestation and whose parents are offered withdrawal of support or do not resuscitate by clinical team for severity of cardiorespiratory illness at or before 12 hours of age)
* newborns diagnosed with congenital heart disease within the first 12 hours of life (presence of a ventricular septum defect and a patent ductus arteriosus is not an exclusion criteria)

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2015-09; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of death and bronchopulmonary dysplasia | 36 weeks post menstrual age

CONTACTS AND LOCATIONS:
Overall Officials: Nitin S Chouthai, MD, Principal Investigator — Wayne State University
Locations (1):
- Hutzel Women's Hospital, Detroit, Michigan, United States